CLINICAL TRIAL: NCT02631070
Title: A Phase 3, Double-blind, Randomized Study to Compare the Efficacy and Safety of Luspatercept (ACE-536) Versus Placebo for the Treatment of Anemia Due to the IPSS-R Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes in Subjects With Ring Sideroblasts Who Require Red Blood Cell Transfusions.
Brief Title: A Study of Luspatercept (ACE-536) to Treat Anemia Due to Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes
Acronym: MEDALIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACE-536-MDS-001; 2015-003454-41 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-12-15 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Luspatercept; Transfusion dependent; Lower risk; Low risk; Myelodysplastic Syndromes; ESA refractory; ESA intolerant; ESA ineligible; ACE-536; Anemia; Ring Sideroblasts; Require Red Blood Cell Transfusions; MEDALIST; MDS; IPSS-R very low/IPSS-R low/IPSS-R intermediate
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm - Luspatercept (ACE-536) (Experimental): Starting dose of 1.0 mg/kg subcutaneous injection every 3 weeks
  Interventions: Drug: Luspatercept
- Control Arm: Placebo (Placebo Comparator): Subcutaneous injection every 3 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Luspatercept
  Other Names: ACE-536
  Arms: Experimental Arm - Luspatercept (ACE-536)
Other: Placebo
  Arms: Control Arm: Placebo

SUMMARY:
The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

This is a Phase 3, double-blind, randomized, placebo-controlled, multicenter study to determine the efficacy and safety of luspatercept (ACE-536) versus placebo in participants with anemia due to the Revised International Prognostic Scoring System (IPSS-R) very low, low, or intermediate MDS with ring sideroblasts who require red blood cell (RBC) transfusions.

DETAILED DESCRIPTION:
Anemia is considered to be one of the most prevalent cytopenias in patients who have myelodysplastic syndromes, an umbrella term used to describe disorders relating to the ineffective production of red blood cells, white blood cells, and/or platelets. Ranging in severity from mild (asymptomatic) to severe, anemia can result in patients requiring regular red blood cell (RBC) transfusions, which can lead to further complications from iron overload. The goal of this study is to assess the safety and efficacy of luspatercept versus placebo in anemic patients who are categorized as International Prognostic Scoring System-Revised (IPSS-R) very low, low, or intermediate risk Myelodysplastic syndrome (MDS), have ring sideroblasts present, and require constant RBC transfusions. The design of the study will allow a period of initial randomization of patients into either the luspatercept or placebo arm, followed by a double-blind treatment period, and then an MDS disease assessment visit. For those patients that are determined to be experiencing clinical benefit as judged from the study Investigator by this disease assessment visit, they will be permitted to enter the double-blind Extension Phase of the study. Once patients are discontinued from study treatment, they will enter a post treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is ≥ 18 years of age the time of signing the informed consent form (ICF).
2. Documented diagnosis of MDS according to World Health Organization (WHO)/French American British (FAB) classification that meets IPSS R classification of very low, low, or intermediate risk disease, and:

Ring sideroblast ≥ 15% of erythroid precursors in bone marrow or ≥ 5% (but < 15%) if SF3B1 mutation is present.

* < 5% blasts in bone marrow
* Peripheral blood white blood cell (WBC) count < 13,000/µL 3. Requires red blood cell RBC transfusions 4. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2 5. Subjects who are refractory/intolerant/ineligible to prior erythropoietin-stimulating agents (ESA) treatment, defined as:
* Refractory to prior - erythropoietin stimulating agents treatment: documentation of non-response or response that is no longer maintained to prior ESA-containing regimen, either as single agent or combination (eg, with granulocyte colony stimulating factor (G-CSF); ESA regimen must have been either recombinant human erythropoietin (rHu EPO) ≥ 40,000 IU/wk for at least 8 doses or equivalent OR darbepoetin alpha ≥ 500 μg Q3W for at least 4 doses or equivalent
* Intolerant to prior ESA treatment: documentation of discontinuation of prior ESA-containing regimen, either as single agent or combination (eg, with G-CSF), at any time after introduction due to intolerance or an adverse event
* ESA ineligible: low chance of response to ESA base on endogenous serum erythropoietin level > 200 U/L for subjects not previously treated with ESAs

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Prior therapy with disease modifying agents for underlying MDS disease.
2. Previously treated with either luspatercept (ACE-536) or sotatercept (ACE-011)
3. MDS associated with del 5q cytogenetic abnormality
4. Secondary MDS, ie, MDS that is known to have arisen as the result of chemical injury or treatment with chemotherapy and/or radiation for other diseases.
5. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding

   - iron deficiency to be determined by serum ferritin less than or equal to 15 ug/L and additional testing if clinically indicated (eg, calculated transferrin saturation [iron/total iron binding capacity less than or equal to 20%] or bone marrow aspirate stain for iron).
6. Prior allogeneic or autologous stem cell transplant
7. Known history of diagnosis of acute myeloid leukemia (AML)
8. Use of any of the following within 5 weeks prior to randomization:

   * anticancer cytotoxic chemotherapeutic agent or treatment
   * corticosteroid, except for subjects on a stable or decreasing dose for ≥ 1 week prior to randomization for medical conditions other than MDS
   * iron-chelating agents, except for subjects on a stable or decreasing dose for at least 8 weeks prior to randomization
   * other RBC hematopoietic growth factors (eg, Interleukin-3)
   * investigational drug or device, or approved therapy for investigational use. If the half-life of the previous investigational product is known, use within 5 times the half-life prior to randomization or within 5 weeks, whichever is longer is excluded.
9. Prior history of malignancies, other than MDS, unless the subject has been free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed:

   * Basal or squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
10. Major surgery within 8 weeks prior to randomization. Subjects must have completely recovered from any previous surgery prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ito, MD, Study Director — Celgene
Locations (74):
- United States (13):
  - Stanford Cancer Center, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Ochsner Medical Institutions, New Orleans, Louisiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia-Presbyterian Medical Center, New York, New York
  - Montefiore Medical Center Albert Einstein Cancer Center, The Bronx, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (7):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - AZ Sint-Jan AV Brugge, Bruges
  - UZ Brussels, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Canada (4):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- France (11):
  - CHU d'Angers, Angers
  - CHU Hotel, Grenoble
  - CHRU de Lille-Hopital Claude Huriez Service des Maladies du Sang, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU de Nice Archet I, Nice
  - Hopital Saint Louis, Paris
  - Hopital Haut Leveque, Pessac
  - Centre hospitalier Lyon Sud Hematologie, Pierre-Bénite
  - Hopital civil, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Hopital Bretonneau, Tours
- Germany (6):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien Hospital, Düsseldorf
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der Technischen Universität München, München
- Italy (8):
  - Azienda Ospedaliera Santi Antonio Biagio E Cesare Arrigo, Allessandria
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico Sorsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Sanitaria Locale Lecce, Lecce
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Fondazione PTV Policlinico Tor Vergata, Roma
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Ziekenhuis, Hoofddorp
- Spain (8):
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario Vall D hebron, Barcelona
  - Instituto Catalan de Oncologia-Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Skanes Universitetssjukhus Lund, Lund
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Turkey (Türkiye) (4):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Ankara University Medical Faculty Cebeci Hospital, Ankara
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- United Kingdom (6):
  - Aberdeen Royal Infirmary, Aberdeen
  - John Radcliffe Hospital, Headington
  - St James University Hospital, Leeds
  - Guys Hospital, London
  - Kings College Hospital, London
  - Kings Mill Hospital, Sutton in Ashfield

REFERENCES:
- [Background] Porter J. Beyond transfusion therapy: new therapies in thalassemia including drugs, alternate donor transplant, and gene therapy. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):361-370. doi: 10.1182/asheducation-2018.1.361. PMID 30504333
- [Background] Piga A, Perrotta S, Gamberini MR, Voskaridou E, Melpignano A, Filosa A, Caruso V, Pietrangelo A, Longo F, Tartaglione I, Borgna-Pignatti C, Zhang X, Laadem A, Sherman ML, Attie KM. Luspatercept improves hemoglobin levels and blood transfusion requirements in a study of patients with beta-thalassemia. Blood. 2019 Mar 21;133(12):1279-1289. doi: 10.1182/blood-2018-10-879247. Epub 2019 Jan 7. PMID 30617198
- [Result] Fenaux P, Platzbecker U, Mufti GJ, Garcia-Manero G, Buckstein R, Santini V, Diez-Campelo M, Finelli C, Cazzola M, Ilhan O, Sekeres MA, Falantes JF, Arrizabalaga B, Salvi F, Giai V, Vyas P, Bowen D, Selleslag D, DeZern AE, Jurcic JG, Germing U, Gotze KS, Quesnel B, Beyne-Rauzy O, Cluzeau T, Voso MT, Mazure D, Vellenga E, Greenberg PL, Hellstrom-Lindberg E, Zeidan AM, Ades L, Verma A, Savona MR, Laadem A, Benzohra A, Zhang J, Rampersad A, Dunshee DR, Linde PG, Sherman ML, Komrokji RS, List AF. Luspatercept in Patients with Lower-Risk Myelodysplastic Syndromes. N Engl J Med. 2020 Jan 9;382(2):140-151. doi: 10.1056/NEJMoa1908892. PMID 31914241
- [Result] Komrokji RS. Luspatercept in Myelodysplastic Syndromes: Who and When? Hematol Oncol Clin North Am. 2020 Apr;34(2):393-400. doi: 10.1016/j.hoc.2019.10.004. Epub 2020 Jan 21. PMID 32089218
- [Result] Fenaux P, Kiladjian JJ, Platzbecker U. Luspatercept for the treatment of anemia in myelodysplastic syndromes and primary myelofibrosis. Blood. 2019 Feb 21;133(8):790-794. doi: 10.1182/blood-2018-11-876888. Epub 2019 Jan 2. PMID 30602619
- [Derived] Germing U, Fenaux P, Platzbecker U, Buckstein R, Santini V, Diez-Campelo M, Yucel A, Tang D, Fabre S, Zhang G, Zoffoli R, Ha X, Miteva D, Hughes C, Komrokji RS, Zeidan AM, Garcia-Manero G. Improved benefit of continuing luspatercept therapy: sub-analysis of patients with lower-risk MDS in the MEDALIST study. Ann Hematol. 2023 Feb;102(2):311-321. doi: 10.1007/s00277-022-05071-8. Epub 2023 Jan 13. PMID 36635381

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 229 participants were randomized and treated.
Groups:
- Luspatercept: Luspatercept 1.0 mg/Kg SC on Day 1 of each 21-day treatment cycle
- Placebo: Placebo (Volume equivalent to experimental arm) SC on Day 1 of each 21-day treatment cycle
Period: Overall Study
Arm/Group | Luspatercept | Placebo
Started | 153 | 76
Completed | 4 | 12
Not Completed | 149 | 64
Not completed — Withdrawal by Subject | 35 | 13
Not completed — Death | 45 | 24
Not completed — Lost to Follow-up | 5 | 1
Not completed — Transition to rollover protocol | 52 | 21
Not completed — Other reasons | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luspatercept | Placebo | Total
Number analyzed (Participants) | 153 | 76 | 229
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (8.68) | 70.7 (10.88) | 70.6 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 26 | 85
  Male | 94 | 50 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 115 | 52 | 167
  Unknown or Not Reported | 35 | 20 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  White | 107 | 51 | 158
  Not Collected or Reported | 44 | 24 | 68
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Achieved Red Blood Cell Transfusion Independence (RBC-TI) ≥ 8 Weeks From Week 1 to Week 24
Description: RBC-TI response was defined as the absence of any Red Blood Cells (RBC) transfusion during any consecutive 56-day (8-week) period (ie, Days 1 to 56, Days 2 to 57, Days 3 to 58, etc.) during the first 24 weeks of study treatment. Participants had to have at least 56 days (≥ 8 weeks) of transfusion independence prior to (and including) the Week 24 cut-off date to qualify as a responder. Participants who failed to achieve RBC-TI at least 56 days prior to or on the cut-off date were counted as non-responders.
Time Frame: From Week 1 through Week 24 of study treatment
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percent of Participants | 37.91 [30.20 to 46.10] | 13.16 [6.49 to 22.87]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Common Risk Difference on Response Rate = 24.56, 95% CI 2-sided [14.48 to 34.64]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.065, 95% CI 2-sided [2.278 to 11.259]

2. Secondary Outcome: Percentage of Participants Who Achieved Red Blood Cell Transfusion Independence (RBC-TI) ≥ 12 Weeks From Week 1 to Week 24
Description: RBC-TI Response was defined as the absence of any Red Blood Cells (RBC) transfusion during any consecutive 84-day (12-week) period (ie, Days 1 to 84, Days 2 to 85, Days 3 to 86, etc.) during the first 24 weeks of treatment.
Time Frame: From Week 1 through Week 24 of study treatment
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percent of Participants | 28.10 [21.14 to 35.93] | 7.89 [2.95 to 16.40]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Common Risk Difference on Response Rate = 20.00, 95% CI 2-sided [10.92 to 29.08]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.071, 95% CI 2-sided [2.002 to 12.844]

3. Secondary Outcome: Percentage of Participants Who Achieved Red Blood Cell Transfusion Independence (RBC-TI) ≥ 12 Weeks From Week 1 to Week 48
Description: RBC-TI Response was defined as the absence of any Red Blood Cells (RBC) transfusion during any consecutive 84-day (12-week) period (ie, Days 1 to 84, Days 2 to 85, Days 3 to 86, etc.) during the first 48 weeks of treatment.
Time Frame: From Week 1 through Week 48 of study treatment
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percent of Participants | 33.33 [25.93 to 41.40] | 11.84 [5.56 to 21.29]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Common Risk Difference on Response Rate = 21.37, 95% CI 2-sided [11.23 to 31.51]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.045, 95% CI 2-sided [1.827 to 8.956]

4. Secondary Outcome: Percentage of Participants Who Achieved Red Blood Cell Transfusion Independence (RBC-TI) ≥ 8 Weeks From Week 1 Through Week 48
Description: RBC-TI response was defined as the absence of any Red Blood Cells (RBC) transfusion during any consecutive 56-day (8-week) period (ie, Days 1 to 56, Days 2 to 57, Days 3 to 58, etc.) during Week 1 through Week 48. Participants had to have at least 56 days (≥ 8 weeks) of transfusion independence prior to (and including) the Week 48 cut-off date to qualify as a responder. Participants who failed to achieve RBC-TI at least 56 days prior to Week 48 were counted as non-responders.
Time Frame: From Week 1 through Week 48 of study treatment
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percentage of Participants | 45.10 [37.05 to 53.34] | 15.79 [8.43 to 25.96]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Common Risk Difference on Response Rate = 29.55, 95% CI 2-sided [18.73 to 40.36]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.306, 95% CI 2-sided [2.526 to 11.146]

5. Secondary Outcome: Change From Baseline in RBC Units Transfused Over Fixed 16-Week Period
Description: Mean change in total number of Red Blood Cells (RBC) units transfused over a fixed 16-week period (Week 9-24 or Week 33-48) from the total number of RBC units transfused in the 16 weeks immediately on or prior to first dose of study treatment.
Time Frame: At Baseline (16 weeks prior to first dose of study treatment) and Weeks 9 to 24 or Weeks 33 to 48
Population: All treated participants with available measurements at the indicated timepoints
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 128 | 68
Units
  Weeks 9 to 24 | -3.0 (5.17) | 0.4 (4.25)
  Weeks 33 to 48: number analyzed (Participants) | 78 | 12
  Weeks 33 to 48 | -4.9 (4.22) | -3.9 (7.14)

6. Secondary Outcome: Percentage of Participants Who Achieved a Modified Hematologic Erythroid Response (mHI-E) Over Any Consecutive 56-Day Period
Description: A modified HI-E response was defined as the percentage of participants meeting the modified HI-E per the International Working Group (IWG) sustained over 56-day consecutive period during the Treatment period. For participants with a baseline RBC transfusion burden of ≥ 4 units/8 weeks, a mHI-E was defined as a reduction in RBC transfusion of at least 4 units/8 weeks; for participants with baseline RBC transfusion burden of <4 units/8 weeks, mHI-E, was defined as a mean increase in hemoglobin of ≥ 1.5 g/dL for 8 weeks in the absence of RBC transfusions.
Time Frame: Week 1 through 24 or Week 1 Through Week 48
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percentage of Participants
  Week 1 Through Week 24 | 52.9 [44.72 to 61.05] | 11.8 [5.56 to 21.29]
  Week 1 Through Week 48 | 58.8 [50.59 to 66.71] | 17.1 [9.43 to 27.47]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Week 1 -24; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Week 1 - 48; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Participants Who Achieved a Mean Hemoglobin (Hgb) Increase of at Least 1.0 g/dL Over Any Consecutive 56-Day Period in Absence of Red Blood Cells (RBC) Transfusions
Description: A mean hgb increase of ≥ 1.0 g/dL was analyzed as the percentage of participants with a hgb increase ≥ 1.0 g/dL compared with baseline (after applying the 14/3 day rule) that was sustained over any consecutive 56-day (8-week) period in the absence of RBC transfusions during the treatment period. (Week 1 through Week 24 and Week 1 through Week 48).
Time Frame: Week 1 though Week 24 and Week 1 through 48
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percentage of Participants
  Week 1 Through Week 24 | 35.3 [27.75 to 43.42] | 7.9 [2.95 to 16.40]
  Week 1 Through Week 48 | 41.2 [33.29 to 49.41] | 10.5 [4.66 to 19.69]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Week 1 Through Week 24; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Week 1 Through Week 48; Test type: Superiority; p < 0.0001, Fisher Exact

8. Secondary Outcome: Duration of Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 24
Description: Duration of RBC-TI was defined as the longest duration of response for participants who achieved RBC-TI of ≥ 8 weeks during the treatment period Week 1 through Week 24. Participants who maintained RBC-TI through the end of the treatment period were censored at the date of IP discontinuation or death, whichever occurred first. Median was estimated from unstratified Kaplan Meier method.
Time Frame: From start of study treatment to 16 weeks after last dose, up to approximately 93 weeks
Population: All treated participants who achieved RBC-TI ≥ 8 weeks during Week 1 through Week 24 of study treatment
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 58 | 10
Weeks | 30.6 [20.6 to 40.6] | 13.6 [9.1 to 54.9]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0445, Log Rank; Hazard Ratio (HR) = 0.446, 95% CI 2-sided [0.196 to 1.013] — HR is from the Cox proportional hazards model

9. Secondary Outcome: Duration of Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 48
Description: Duration of RBC-TI was defined as the longest duration of response for participants who achieved RBC-TI of ≥ 8 weeks during the treatment period Week 1 through Week 48. Participants who maintained RBC-TI through the end of the treatment period were censored at the date of IP discontinuation or death, whichever occurred first. Median was estimated from unstratified Kaplan Meier method.
Time Frame: From start of study treatment to 16 weeks after last dose, up to approximately 93 weeks
Population: All treated participants who achieved RBC-TI ≥ 8 weeks during Week 1 through Week 48 of study treatment
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 69 | 12
Weeks | 30.6 [20.6 to 50.9] | 18.6 [10.9 to NA] — Upper limit could not be estimated due to insufficient number of events
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.5121, Log Rank; Hazard Ratio (HR) = 0.784, 95% CI 2-sided [0.362 to 1.699] — HR is from the Cox proportional hazards model

10. Secondary Outcome: Mean Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Global Quality of Life Score
Description: The EORTC questionnaire is a validated health-related quality of life (HRQoL) measure applicable to participants with any cancer diagnosis. Version 3.0 of the questionnaire was used in the study.
  It is composed of 30 items that address 15 domains, including one global health status, functional domains, and symptom domains. Domain scores are transformed to a 0 to 100 scale, where higher scores on the global quality of life score indicate better function. As such, a positive change from Baseline score indicates an improvement in quality of life.
Time Frame: Baseline and Cycle 3, Day 1 (C3 D1), C5 D1, C7 D1, Week 25, every other cycle during extension phase (C1 D1, C3 D1, C5 D1, etc. up to C59 D1) and end of treatment. Each cycle is composed of 21 days.
Population: All treated participants who completed the EORTC QLQ-C30 assessment at baseline and at least one post-baseline assessment visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 149 | 76
Score on a scale
  Cycle 3 Day 1 (C3 D1): number analyzed (Participants) | 133 | 69
  Cycle 3 Day 1 (C3 D1) | -4.1 (21.01) | 0.1 (15.95)
  C5 D1: number analyzed (Participants) | 129 | 65
  C5 D1 | -2.4 (20.73) | 2.2 (17.13)
  C7 D1: number analyzed (Participants) | 108 | 59
  C7 D1 | -2.1 (23.04) | -0.6 (18.63)
  Week 25: number analyzed (Participants) | 110 | 53
  Week 25 | -1.8 (21.75) | 0.2 (18.88)
  Extension Phase C1 D1: number analyzed (Participants) | 48 | 8
  Extension Phase C1 D1 | 0.0 (25.32) | 6.3 (14.60)
  Extension Phase C3 D1: number analyzed (Participants) | 83 | 17
  Extension Phase C3 D1 | 2.0 (19.68) | -3.9 (26.86)
  Extension Phase C5 D1: number analyzed (Participants) | 77 | 15
  Extension Phase C5 D1 | 0.8 (18.40) | 0.6 (20.04)
  Extension Phase C7 D1: number analyzed (Participants) | 74 | 13
  Extension Phase C7 D1 | -0.5 (20.03) | 3.8 (20.87)
  Extension Phase C9 D1: number analyzed (Participants) | 69 | 7
  Extension Phase C9 D1 | -2.4 (18.42) | 11.9 (19.75)
  Extension Phase C11 D1: number analyzed (Participants) | 60 | 7
  Extension Phase C11 D1 | -1.8 (19.53) | 4.8 (24.47)
  Extension Phase C13 D1: number analyzed (Participants) | 58 | 6
  Extension Phase C13 D1 | -2.6 (20.84) | 8.3 (24.15)
  Extension Phase C15 D1: number analyzed (Participants) | 57 | 6
  Extension Phase C15 D1 | 3.1 (18.27) | 4.2 (27.26)
  Extension Phase C17 D1: number analyzed (Participants) | 55 | 3
  Extension Phase C17 D1 | -0.6 (19.03) | 13.9 (26.79)
  Extension Phase C19 D1: number analyzed (Participants) | 51 | 3
  Extension Phase C19 D1 | -1.6 (18.78) | -16.7 (14.43)
  Extension Phase C21 D1: number analyzed (Participants) | 45 | 2
  Extension Phase C21 D1 | 3.1 (18.32) | 4.2 (17.68)
  Extension Phase C23 D1: number analyzed (Participants) | 38 | 1
  Extension Phase C23 D1 | 0.9 (17.84) | 16.7 (NA) — No standard deviation could be determined because a single participant was analyzed
  Extension Phase C25 D1: number analyzed (Participants) | 37 | 1
  Extension Phase C25 D1 | -2.0 (18.15) | 16.7 (NA) — No standard deviation could be determined because a single participant was analyzed
  Extension Phase C27 D1: number analyzed (Participants) | 37 | 0
  Extension Phase C27 D1 | 2.5 (20.40) |
  Extension Phase C29 D1: number analyzed (Participants) | 36 | 0
  Extension Phase C29 D1 | 2.1 (21.12) |
  Extension Phase C31 D1: number analyzed (Participants) | 33 | 0
  Extension Phase C31 D1 | -0.3 (15.93) |
  Extension Phase C33 D1: number analyzed (Participants) | 34 | 0
  Extension Phase C33 D1 | -1.5 (19.41) |
  Extension Phase C35 D1: number analyzed (Participants) | 30 | 0
  Extension Phase C35 D1 | 3.6 (23.33) |
  Extension Phase C37 D1: number analyzed (Participants) | 31 | 0
  Extension Phase C37 D1 | 0.5 (22.04) |
  Extension Phase C39 D1: number analyzed (Participants) | 26 | 0
  Extension Phase C39 D1 | 0.3 (23.63) |
  Extension Phase C41 D1: number analyzed (Participants) | 24 | 0
  Extension Phase C41 D1 | 6.6 (20.11) |
  Extension Phase C43 D1: number analyzed (Participants) | 19 | 0
  Extension Phase C43 D1 | 4.8 (15.29) |
  Extension Phase C45 D1: number analyzed (Participants) | 15 | 0
  Extension Phase C45 D1 | -2.2 (21.24) |
  Extension Phase C47 D1: number analyzed (Participants) | 12 | 0
  Extension Phase C47 D1 | 1.4 (19.08) |
  Extension Phase C49 D1: number analyzed (Participants) | 11 | 0
  Extension Phase C49 D1 | -3.8 (16.40) |
  Extension Phase C51 D1: number analyzed (Participants) | 3 | 0
  Extension Phase C51 D1 | 8.3 (8.33) |
  Extension Phase C53 D1: number analyzed (Participants) | 4 | 0
  Extension Phase C53 D1 | 12.5 (10.76) |
  Extension Phase C55 D1: number analyzed (Participants) | 3 | 0
  Extension Phase C55 D1 | 2.8 (17.35) |
  Extension Phase C57 D1: number analyzed (Participants) | 2 | 0
  Extension Phase C57 D1 | 12.5 (5.89) |
  Extension Phase C59 D1: number analyzed (Participants) | 1 | 0
  Extension Phase C59 D1 | 16.7 (NA) — No standard deviation could be determined because a single participant was analyzed |
  End of Treatment: number analyzed (Participants) | 88 | 33
  End of Treatment | -9.2 (23.97) | -0.8 (23.07)

11. Secondary Outcome: Percentage of Participants Who Achieved a Hematologic Improvement in Neutrophil Response (HI-N) Over Any Consecutive 56-day Period
Description: Percentage of participants who achieved a hematologic improvement in neutrophil response (HI-N) per IWG criteria sustained over any consecutive 56-day (8-week) period, during the treatment period (Week 1 to Week 24 and Week 1 to Week 48) HI-N was defined as at least a 100% increase and an absolute increase > 0.5 X 10^9/L.
Time Frame: Week 1 through Week 24 or Week 1 Through Week 48 of study treatment
Population: All treated participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 15 | 10
Percentage of Participants
  Week 1 Through Week 24 | 13.3 [1.66 to 40.46] | 0 [0.00 to 30.85]
  Week 1 Through Week 48 | 20.0 [4.33 to 48.09] | 10.0 [0.25 to 44.50]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Week 1 -24; Test type: Superiority; p = 0.2382, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Week 1 - 48; Test type: Superiority; p = 0.5127, Cochran-Mantel-Haenszel

12. Secondary Outcome: Percentage of Participants Who Achieved a Hematologic Improvement in Platelet Response (HI-P) Over Any Consecutive 56-day Period
Description: Percentage of participants who achieved a hematologic improvement platelet response (HI-P) was defined as the percentage of participants meeting the HI-P criteria per the IWG sustained over any consecutive 56-day (8-week) period (Week 1 to Week 24 and Week 1 to Week 48) during the treatment period. HI - P reponse was defined as:
  * Absolute increase of ≥ 30 X 10^9/L in platelets for participants starting with > 20 X 10^9/L platelets
  * Increase in platelets from < 20 X 10^9/L to > 20 X 10^9/L and by at least 100%
Time Frame: Week 1 through Week 24 or Week 1 Through Week 48 of study treatment
Population: All treated participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 8 | 6
Percentage of Participants
  Week 1 Through Week 24 | 50.0 [15.70 to 84.30] | 33.3 [4.33 to 77.72]
  Week 1 Through Week 48 | 62.5 [24.49 to 91.48] | 33.3 [4.33 to 77.72]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Week 1 -24; Test type: Superiority; p = 0.5479, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Week 1 - 48; Test type: Superiority; p = 0.2980, Cochran-Mantel-Haenszel

13. Secondary Outcome: Change From Baseline in Mean Serum Ferritin
Description: Mean change from baseline in mean serum ferritin was calculated as the difference of postbaseline mean serum ferritin (averaged over the specified timepoints) and baseline mean serum ferritin.
Time Frame: Baseline and Week 9 through Week 24 and Week 33 through Week 48
Population: All treated participants with available measurements
Measure: Least Squares Mean (Standard Error); unit: ug/L
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 148 | 74
ug/L
  Weeks 9-24 | -2.7 (54.05) | 226.5 (68.02)
  Weeks 33-48: number analyzed (Participants) | 89 | 16
  Weeks 33-48 | -72.0 (74.76) | 247.4 (140.96)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Week 9 Through 24; Test type: Superiority; p = 0.0024, ANCOVA; LS Mean Difference = -229.1, 95% CI 2-sided [-375.8 to -82.4], Standard Error of Mean 74.43
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Week 33 Through 48; Test type: Superiority; p = 0.0294, ANCOVA; LS Mean Difference = -319.5, 95% CI 2-sided [-606.3 to -32.7], Standard Error of Mean 144.57

14. Secondary Outcome: Change From Baseline in Mean Daily Dose of Iron Chelation Therapy (ICT)
Description: Mean change from baseline in mean daily dose of ICT averaged over Week 9 to Week 24 or Week 33 to Week 48. For each participant, the mean change in daily dose of ICT was calculated as the difference of postbaseline mean daily dose and baseline mean daily dose.
Time Frame: Baseline and Week 9 through Week 24 and Week 33 through Week 48 of study treatment
Population: All treated participants with available measurements
Measure: Least Squares Mean (Standard Error); unit: mg/day
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 128 | 68
mg/day
  Weeks 9-24 | 10.0 (29.25) | 51.0 (35.92)
  Weeks 33-48: number analyzed (Participants) | 78 | 12
  Weeks 33-48 | -148.8 (46.13) | -123.8 (92.19)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Weeks 9 Through 24; Test type: Superiority; p = 0.3087, ANCOVA; LS Mean Difference = -41.0, 95% CI 2-sided [-120.3 to 38.2], Standard Error of Mean 40.18
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Weeks 33 Through 48; Test type: Superiority; p = 0.7903, ANCOVA; LS Mean Difference = -24.9, 95% CI 2-sided [-210.7 to 160.8], Standard Error of Mean 93.42

15. Secondary Outcome: Time to Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 24
Description: Time to RBC-TI was defined as the time between first dose date and the date of onset of RBC-TI first observed for participants who achieved RBC-TI of ≥ 8 weeks during Week 1 through Week 24
Time Frame: From first dose to Week 24 of study treatment
Population: All participants who achieved RBC-TI ≥ 8 weeks during Week 1 through Week 24
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 58 | 10
Days | 17.2 (29.40) | 26.0 (31.83)

16. Secondary Outcome: Time to Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 48
Description: Time to RBC-TI was defined as the time between first dose date and the date of onset of RBC-TI first observed for participants who achieved RBC-TI of ≥ 8 weeks during Week 1 through Week 48
Time Frame: From first dose to Week 48 of study treatment
Population: All participants who achieved RBC-TI ≥ 8 weeks during Week 1 through Week 48
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 69 | 12
Days | 40.3 (61.03) | 57.2 (79.18)

17. Secondary Outcome: Percentage of Participants Who Progressed to Acute Myeloid Leukemia (AML)
Description: Percentage of participants progressing to AML throughout the course of the study
Time Frame: From randomization to study completion (up to approximately 57 months)
Population: All treated participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Percentage of Participants | 2.6 | 3.9

18. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Progression
Description: Time to AML progression was defined as the time between randomization date and the first diagnosis of AML as per World Health Organization (WHO) classification of ≥ 20% blasts in peripheral blood or bone marrow. Participants with a diagnosis of AML were considered to have had an event, participants who did not progress to AML at the time of analysis were censored at the last assessment date which did not indicate progression to AML.
Time Frame: From randomization to study completion (up to approximately 57 months)
Population: All treated participants who progressed to AML
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 4 | 3
Months | NA [NA to NA] — Median was not estimable due to the insufficient number of events | NA [NA to NA] — Median was not estimable due to the insufficient number of events

19. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from the date of study drug randomization to death due to any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for those who discontinued from the study or were lost to follow-up.
Time Frame: From randomization to study completion (up to approximately 57 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Months | 46.0 [42.0 to NA] — Upper limit could not be estimated because of the insufficient number of events | NA [43.1 to NA] — Median and Upper limit could not be estimated because of the insufficient number of events
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.9580, Log Rank; Hazard Ratio (HR) = 0.986, 95% CI 2-sided [0.595 to 1.636] — HR is from the Cox proportional hazards model

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: The outcome measure describes the number of participants who experienced different types of Treatment-emergent adverse events (TEAEs).
  TEAEs were defined as Adverse Events (AEs) that started on or after the day of the first dose and on or before 42 days after the last dose of IP.
  The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event. The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: From date of first dose up to 42 days after the last dose (up to approximately 83 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Participants
  ≥ 1 TEAE | 151 | 70
  ≥ 1 Suspected Related TEAE | 71 | 26
  ≥ 1 Serious TEAE | 66 | 23
  ≥ 1 Suspected Related Serious TEAE | 6 | 0
  ≥ 1 TEAE CTCAE Toxicity Grade (GR) 5 | 8 | 4
  ≥ 1 Suspected Related TEAE With CTCAE GR 5 | 0 | 0
  ≥ 1 TEAE with CTCAE GR 3 or 4 | 86 | 34
  ≥ 1 Suspected Related TEAE With CTCAE GR 3 or 4 | 13 | 3
  ≥ 1 TEAE Leading to Dose Interruption | 42 | 4
  ≥ 1 TEAE Leading to Dose Reduction | 9 | 0
  ≥ 1 TEAE Leading to Study Drug Discontinuation | 22 | 6

21. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Apparent Clearance (CL/F)
Description: Apparent total plasma clearance was calculated as Dose/Area Under the Curve to infinity (ꝏ).
Time Frame: Blood serum samples taken pre-dose at Cycle 1 Day 1 (C1, D1), C1 D8, C1 D15, C2 D1, C4 D1, C5 D8, C6 D1 and Week 25 visit, extension phase C4 D1 and Day 1 of every fourth treatment cycle thereafter.
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of luspatercept and had measurable luspatercept serum concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
L/day | 0.516 (41.2) |

22. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Apparent Volume of Distribution of the Central Compartment (V1/F)
Description: Apparent volume of distribution of luspatercept was calculated according to the equation Vz = (CL)/λ.
Time Frame: as for outcome 21
Population: Pharmacokinetic population included all participants who received at least 1 dose of luspatercept and had measurable luspatercept serum concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
L | 9.68 (26.5) |

23. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Elimination Half-life (t1/2)
Description: Terminal phase half-life was calculated according to the following equation: t1/2 = 0.693/λz.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
Day | 13.0 (31.6) |

24. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Time to Reach Maximum Concentration (Tmax)
Description: Tmax was defined as the observed time to maximum plasma concentration of luspatercept.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Median (Full Range); unit: Day
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
Day | 5.40 [3.12 to 6.69] |

25. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Maximum Concentration for the First Dose (Cmax)
Description: Cmax was defined as the observed maximum plasma concentration, obtained directly from the observed concentration versus time.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
μg/mL | 5.77 (20.5) |

26. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Maximum Concentration for the Starting Dose (Cmax) at Steady State
Description: Cmax was defined as the observed maximum plasma concentration, obtained directly from the observed concentration at a steady state.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
μg/mL | 9.17 (29.9) |

27. Secondary Outcome: Pharmacokinetic (PK) Parameters: Bayesian Estimate of Maximum Concentration for the Area Under the Curve at Steady State for Starting Dose (AUC^ss)
Description: Area under the curve steady state was defined as the area under the plasma concentration-time curve for a steady state. calculated by the linear trapezoidal rule.
Time Frame: as for outcome 21
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day/μg/mL
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 0
day/μg/mL | 145 (38.3) |

28. Secondary Outcome: Participants With Pre-Existing and/or Treatment-Emergent Antidrug Antibodies (ADA)
Description: Number of participants with positive ADA prior to taking study drug and/or during study. A participant was counted as "treatment-emergent" if there was a positive post-baseline sample while the baseline sample was ADA negative, or there was a positive post-baseline sample with a titer ≥ 4-fold of the baseline titer while the baseline sample was ADA positive. A participant was counted as "preexisting" if the baseline sample was ADA positive and the participant was not qualified for "treatment-emergent."
Time Frame: From randomization to 1 year post first dose
Population: Safety population of participants with ADA samples collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 153 | 76
Participants
  Pre-Existing ADA | 7 | 2
  Treatment Emergent ADA | 11 | 3
  Treatment Emergent Neutralizing ADA | 5 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to approximately 57 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 91 weeks)
Arm/Group | Luspatercept | Placebo
All-Cause Mortality (participants affected / at risk) | 45/153 | 24/76
Serious Adverse Events (participants affected / at risk) | 66/153 | 23/76
Other Adverse Events (participants affected / at risk) | 145/153 | 63/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=153) | Placebo (N=76)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 3 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 2
Pneumonia moraxella (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 1
Septic shock (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 3
Femur fracture (Injury, poisoning and procedural complications) | 6 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic bone injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Systemic mastocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Thrombosis in device (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=153) | Placebo (N=76)
Anaemia (Blood and lymphatic system disorders) | 14 | 6
Neutropenia (Blood and lymphatic system disorders) | 8 | 7
Palpitations (Cardiac disorders) | 11 | 5
Tachycardia (Cardiac disorders) | 8 | 0
Vertigo (Ear and labyrinth disorders) | 12 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 4
Abdominal pain upper (Gastrointestinal disorders) | 11 | 2
Constipation (Gastrointestinal disorders) | 21 | 7
Diarrhoea (Gastrointestinal disorders) | 44 | 8
Nausea (Gastrointestinal disorders) | 35 | 6
Vomiting (Gastrointestinal disorders) | 14 | 5
Asthenia (General disorders) | 40 | 9
Fatigue (General disorders) | 46 | 11
Influenza like illness (General disorders) | 9 | 3
Malaise (General disorders) | 8 | 3
Oedema peripheral (General disorders) | 37 | 13
Pyrexia (General disorders) | 19 | 6
Bronchitis (Infections and infestations) | 19 | 1
Influenza (Infections and infestations) | 11 | 0
Nasopharyngitis (Infections and infestations) | 18 | 4
Upper respiratory tract infection (Infections and infestations) | 19 | 4
Urinary tract infection (Infections and infestations) | 21 | 4
Fall (Injury, poisoning and procedural complications) | 25 | 7
Alanine aminotransferase increased (Investigations) | 9 | 3
Aspartate aminotransferase increased (Investigations) | 10 | 1
Weight decreased (Investigations) | 9 | 5
Decreased appetite (Metabolism and nutrition disorders) | 14 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 2
Iron overload (Metabolism and nutrition disorders) | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Dizziness (Nervous system disorders) | 35 | 4
Headache (Nervous system disorders) | 27 | 5
Syncope (Nervous system disorders) | 10 | 1
Anxiety (Psychiatric disorders) | 9 | 1
Confusional state (Psychiatric disorders) | 9 | 0
Depression (Psychiatric disorders) | 9 | 5
Insomnia (Psychiatric disorders) | 13 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 3
Hypertension (Vascular disorders) | 16 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT02631070/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT02631070/SAP_001.pdf